CLINICAL TRIAL: NCT06583525
Title: Evaluation of the Transition to Adult Care (TAC) Program for High-Risk Youth with Multimorbidity or Rare Disease: a Prospective Observation Cohort Study
Brief Title: Evaluation of the TAC Program
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Alene Toulany, Principal investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000081574
Record Dates: First submitted 2024-08-29; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Youth with Multimorbidity or Rare Dieases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Other: Intensive Transition Support

INTERVENTIONS:
Other: Intensive Transition Support — A multidisciplinary transition team (nurse practitioner and social worker) will coordinate the transition process for each patient across multiple settings, focused on the youth's highest priority needs while also supporting the caregivers. Participants will receive case management and care navigation using an intensive transition support model provided through the partnership of a transition team. The transition team will collaborate with the participants existing care team to help coordinate care, provide consultation, and support adult and primary care accepting these youth for 1 year following the transfer. This Intervention is modelled on best practices by Health Quality Ontario's Quality Standards for Transition from Youth to Adult Health Care Services to support youth at high risk of having poor transitional outcomes as they move from pediatric to adult care.

SUMMARY:
This is a mixed-methods evaluative study examining the effectiveness of the Transition to Adult Care Program at the Hospital for Sick Children (TAC) Program on high-risk youth with medical and psychosocial complexity transitioning to adult and/or primary care services.

The overarching aim is to study the effectiveness of a new interdisciplinary and holistic Transition to Adult Care Program (TAC) on health-related outcomes for high-risk youth with multimorbidity or rare diseases and their caregivers by:

1. Assess the effect of the TAC program on the youth's transition readiness, self-efficacy, self-management, health-related quality of life, and satisfaction.
2. Assess the effect of the TAC program on the caregiver's satisfaction.
3. Explore the experiences, perceptions, needs, and priorities of youth and caregivers participating in the TAC program using qualitative research methods.
4. Describe the feasibility of the TAC program (defined as success in patient recruitment, attendance, participation, retention and transfer).

ELIGIBILITY:
Inclusion Criteria:

Aged 16-18 years old and have a complex medical history, as defined by:

1. Clinical Characteristics: Multi-morbidity (≥ 3 long-term chronic physical and/or mental health conditions (with primary condition being a physical health condition AND/OR Rare disease/ genetic condition.
2. High Risk: No clearly identified adult provider/services following transfer AND/OR experiencing significant barriers related to Social and Structural Determinants of Health.

Exclusion Criteria:

1. Moderate to severe developmental/intellectual disabilities
2. Followed by services at SickKids which has an established transition program/provider
3. Does not provide consent

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Early Identification and Transition Readiness | Baseline,12 months and 24 months
  The change in the patients demonstration of their self-management skills and transition readiness will be assessed using the Transition Readiness Assessment Questionnaire (20-item survey). A scoring of 4 or more across all domains is considered an indicator of transition readiness.
Early Identification and Transition Readiness | Baseline,12 months and 24 months
  The change in the patients self-efficacy in their ability to manage their health and demonstrate transition readiness will be assessed using the General Self-Efficacy Scale (10 item survey). A total score is achieved from a range of 10 to 40, with high scores as an indication of better perceived general self-efficacy.
Early Identification and Transition Readiness | Baseline,12 months and 24 months
  The change in the patients knowledge and confidence in their ability to manage their health and demonstrate transition readiness will be assessed using the Patient Activation Measure (10-item survey). An average net 6-point score increase demonstrating improvement
Early Identification and Transition Readiness - Service Satisfaction | Baseline,12 months and 24 months
  The change in the patients and caregivers satisfaction with transitional health care services will be measured using the Larsen Client Satisfaction Questionnaire (8-item survey).
Information Sharing and Support | 6 to 24 months
  The transition intervention will include providing the patients and caregivers with information on available needs-based services and support. The number of patients who receive this intervention will be assessed via report in the patients medical record.
Information Sharing and Support | 6 to 24 months
  The transition intervention will include offering support from the time of discharge from pediatric services until the first appointment with adult services. The number of patients who receive this intervention will be assessed via report in the patients medical record.
Transition Plan | 6 to 24 months
  The transition intervention will include the co-creating an individualized transition plan to identify the patients transition goals and set timelines. The number of patients who receive this intervention will be assessed via report in the patients medical record.
Coordinated Transition | 6 to 24 months
  The transition intervention will include developing a patient-specific transfer package. The number of patients who receive this intervention will be assessed via report in the patients medical record.
Introduction to Adult Services | 24 to 36 months
  A joint clinic visit will be facilitated by the transition team with the identified receiving adult care provider. The number of patients who have received a warm handover visit with the transition team, primary care provider/service team, will be assessed via report in the patients medical record.
Transition Completion | 24 to 36 months
  Successful transfer will be measured by the attendance of the first appointment with a primary care and/or subspecialty adult care provider between the first 6 to 12 months of transfer from the pediatric provider.
Health-Related Quality of Life | Baseline, 12 months and 24 months
  The change in the patients quality of life will be measured using the The Pediatric Quality of Life Inventory 4.0 Generic Core Scale Teen Report The 23-item survey will assess four core health dimensions (physical functioning, emotional functioning, social functioning and school functioning) transformed into total scores ranging from 0 to 100. An increase in 12 and 24 months follow-up scores from baseline will be measured.
Experience in the process | 24 to 36 months
  Semi-structured qualitative interviews will be conducted with a subset of participants to explore participants; experiences working with the transition team, and satisfaction with the tools and resources used.

SECONDARY OUTCOMES:
Program Feasibility | 24 to 36 months
  The successful implementation of the intervention will be evaluated by assessing the feasibility of the program. The percentage of attended appointments, completed questionnaires, individualized transition plans created, warm handovers completed prior to participants' 18th birthday, and additional clinic visits required will be documented for each participant.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children (SickKids), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No